CLINICAL TRIAL: NCT05811741
Title: Evaluating the Influence of Mandibular Canal Trajectory on the Duration of Postoperative Paresthesia in Patients Undergoing Inferior Alveolar Nerve Lateralization: A Prospective Cohort Study
Brief Title: Impact of Mandibular Canal Trajectory on Paresthesia After Inferior Alveolar Nerve Lateralization
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MUDHF_FB_006
Record Dates: First submitted 2023-04-01; First posted 2023-04-13 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Alveolar Bone Loss; Neurosensory Disorder
Keywords: Mandibular canal; Paresthesia; Dental implants; Survival analysis; Inferior alveolar nerve lateralization
MeSH Terms: conditions — Alveolar Bone Loss; Sensation Disorders; Paresthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study aims to investigate the relationship between mandibular canal trajectory and the duration of postoperative paresthesia in patients undergoing inferior alveolar nerve lateralization. The study will assess mandibular canal trajectory using anatomic factors and evaluate nerve sensory function using subjective and objective tests. Implant success criteria will also be assessed. The study will be conducted on patients who underwent IANL due to mandibular atrophy and were unable to receive standard or short implant placement. Data will be collected at regular follow-up visits up to 1-year post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophied posterior mandible with less than or equal to 6 mm of bone over the inferior alveolar canal
* No previous grafting or implant surgery at the site where nerve lateralization is planned
* No neurosensory impairment
* No contra-indications for implant surgery

Exclusion Criteria:

* Patients who have undergone radiotherapy in the associated area
* Patients using bone-modifying agents
* Smokers with daily consumption of more than ten cigarettes
* Patients with neurosensory impairment due to trauma, tumor, or cancer

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of consecutive patients who were treated with inferior alveolar nerve lateralization (IANL) at Marmara University Faculty of Dentistry between June 2016 and December 2022. The patients had missing teeth in the posterior region of the mandible, in whom standard or short implant placement was not possible due to mandibular atrophy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Light touch test results | Visits at 10 days, 1 month, 2 months, 3 months, 6 months, and 1 year after surgery
  The light touch test is a common diagnostic tool used to assess sensory perception. Patients' lower lip and chin areas will be gently stroked with a soft object, such as a piece of cotton or a brush. The patients will then be asked to report their sensation. If they feel the touch, the response is considered normal. However, any reported changes, such as numbness or tingling, can indicate possible nerve damage or recovery after surgery.
2-point discrimination test results | isits at 10 days, 1 month, 2 months, 3 months, 6 months, and 1 year after surgery.
  The 2-point discrimination test is a neurological examination used to measure tactile spatial acuity. Two points of a caliper will be applied to the patients' lower lip and chin areas. The distance at which a patient can no longer differentiate between the two points provides an indicator of sensory nerve function. Any reported changes in the ability to distinguish between two points may suggest alterations in nerve sensitivity or recovery after surgery.

SECONDARY OUTCOMES:
Thickness of the buccal cortex | At baseline
  This outcome measure evaluates the thickness of the buccal cortex using radiographic measurements obtained from CBCT scans.
Thickness of the mandibular inferior border | At baseline
  This outcome measure evaluates the thickness of the mandibular inferior border using radiographic measurements obtained from CBCT scans.
Diameter of the nerve canal | At baseline
  This outcome measure evaluates the diameter of the nerve canal using radiographic measurements obtained from CBCT scans.
Distance from the nerve canal to the buccal cortex | At baseline
  This outcome measure evaluates the distance from the nerve canal to the buccal cortex using radiographic measurements obtained from CBCT scans.
Distance from the nerve canal to the inferior border of the mandible | At baseline
  This outcome measure evaluates the distance from the nerve canal to the inferior border of the mandible using radiographic measurements obtained from CBCT scans.
Change in Implant stability quotient (ISQ) values: | During implant placement and follow-up visits at 3 months.
  The Implant Stability Quotient (ISQ) is a metric ranging from 1 to 100 that is used to assess implant stability within the bone, with higher values indicating greater stability. To determine ISQ values, resonance frequency analysis (RFA) or sound waves are passed through a specialized peg attached to the implant.
Change in peri-implant bone resorption | At 3 months, and 12 months after surgery.
  This outcome measure evaluates peri-implant bone resorption using OPTG. The amount of bone loss around the implant will be assessed and recorded.
Patient satisfaction | At 12 month follow-up visit
  This outcome measure assesses patient satisfaction using a visual analog scale. Patients will be asked to rate their satisfaction with the treatment outcome at the 12-month follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung RE, Al-Nawas B, Araujo M, Avila-Ortiz G, Barter S, Brodala N, Chappuis V, Chen B, De Souza A, Almeida RF, Fickl S, Finelle G, Ganeles J, Gholami H, Hammerle C, Jensen S, Jokstad A, Katsuyama H, Kleinheinz J, Kunavisarut C, Mardas N, Monje A, Papaspyridakos P, Payer M, Schiegnitz E, Smeets R, Stefanini M, Ten Bruggenkate C, Vazouras K, Weber HP, Weingart D, Windisch P. Group 1 ITI Consensus Report: The influence of implant length and design and medications on clinical and patient-reported outcomes. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:69-77. doi: 10.1111/clr.13342. PMID 30328189
- [Background] Alling CC. Lateral repositioning of inferior alveolar neurovascular bundle. J Oral Surg. 1977 May;35(5):419. No abstract available. PMID 265383
- [Background] Jensen O, Nock D. Inferior alveolar nerve repositioning in conjunction with placement of osseointegrated implants: a case report. Oral Surg Oral Med Oral Pathol. 1987 Mar;63(3):263-8. doi: 10.1016/0030-4220(87)90187-3. PMID 3473351
- [Background] Lorean A, Kablan F, Mazor Z, Mijiritsky E, Russe P, Barbu H, Levin L. Inferior alveolar nerve transposition and reposition for dental implant placement in edentulous or partially edentulous mandibles: a multicenter retrospective study. Int J Oral Maxillofac Surg. 2013 May;42(5):656-9. doi: 10.1016/j.ijom.2013.01.020. Epub 2013 Mar 6. PMID 23481542
- [Background] Palacio Garcia-Ochoa A, Perez-Gonzalez F, Negrillo Moreno A, Sanchez-Labrador L, Cortes-Breton Brinkmann J, Martinez-Gonzalez JM, Lopez-Quiles Martinez J. Complications associated with inferior alveolar nerve reposition technique for simultaneous implant-based rehabilitation of atrophic mandibles. A systematic literature review. J Stomatol Oral Maxillofac Surg. 2020 Sep;121(4):390-396. doi: 10.1016/j.jormas.2019.12.010. Epub 2020 Jan 2. PMID 31904530
- [Background] Kan JY, Lozada JL, Goodacre CJ, Davis WH, Hanisch O. Endosseous implant placement in conjunction with inferior alveolar nerve transposition: an evaluation of neurosensory disturbance. Int J Oral Maxillofac Implants. 1997 Jul-Aug;12(4):463-71. PMID 9274075
- [Background] Abayev B, Juodzbalys G. Inferior Alveolar Nerve Lateralization and Transposition for Dental Implant Placement. Part II: a Systematic Review of Neurosensory Complications. J Oral Maxillofac Res. 2015 Mar 30;6(1):e3. doi: 10.5037/jomr.2014.6103. eCollection 2015 Jan-Mar. PMID 25937874
- [Background] Lee JH, Son YJ, Hwang JH, Baek SH, Jeon JH. Influence of anatomic position and intraoperative exposure of the inferior alveolar nerve on neurosensory disturbance after sagittal split ramus osteotomy: a three-dimensional computed tomography study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Sep;122(3):300-5. doi: 10.1016/j.oooo.2016.04.008. Epub 2016 Apr 23. PMID 27373586
- [Background] Rathod M, Kshirsagar RA, Joshi S, Pawar S, Tapadiya V, Gupta S, Mahajan V. Evaluation of Neurosensory Function Following Inferior Alveolar Nerve Lateralization for Implant Placement. J Maxillofac Oral Surg. 2019 Jun;18(2):273-279. doi: 10.1007/s12663-018-1124-1. Epub 2018 Jun 2. PMID 30996551
- [Background] Zarb GA, Albrektsson T. Consensus report: towards optimized treatment outcomes for dental implants. J Prosthet Dent. 1998 Dec;80(6):641. doi: 10.1016/s0022-3913(98)70048-4. No abstract available. PMID 9830066